CLINICAL TRIAL: NCT01996696
Title: Prevention of Metabolic Syndrome and Increased Weight Using Metformin Concurrent to Androgen Deprivation Therapy and Radiotherapy for Locally Advanced Adenocarcinoma of the Prostate
Acronym: PREMIUM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Results of interim analysis indicate no statistically significant difference in the primary objective between the two arms at baseline and 12 months of follow-up.
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCI-Usmani-01
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Prostatic Neoplasm
Keywords: metformin; metabolic syndrome; weight gain
MeSH Terms: conditions — Prostatic Neoplasms; Metabolic Syndrome; Weight Gain | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Metformin 500 mg PO TID x 30-36 months
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Identical placebo TID x 30-36 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 500 mg PO TID x 30-36 months
  Other Names: Fortamet; Glucophage; Glucophage XR; Glumetza; Riomet
  Arms: Metformin
Drug: Placebo — Identical placebo TID x 30-36 months
  Arms: Placebo

SUMMARY:
In current clinical practice, an acceptable standard treatment for locally advanced prostate cancer is radiation therapy in combination with hormone therapy (called Treatment B or Group B in this study). However, despite our best treatments, there is a risk that the prostate cancer may eventually return. As well, the hormonal therapy that is given to treat the prostate cancer is known to cause some harmful effects, with some patients using the hormones gaining weight, developing diabetes, having increased cholesterol levels, having increased blood pressure, and/or heart problems.

This study is looking at whether Metformin, a drug that is commonly used to treat diabetes, can prevent patients from developing some of the harmful effects of the hormonal therapy. In treating diabetes, Metformin is known to decrease patients' sugar levels and also prevents patients from gaining weight, decreases their cholesterol levels, decreases the number of heart problems and allows patients to live longer. As a result, the researchers in this study are hopeful that Metformin will also be beneficial for men with prostate cancer on hormonal therapy by preventing them from developing these problems.

DETAILED DESCRIPTION:
This study will examine the role of Metformin as a means to prevent increases in weight as well as the prevalence and severity of metabolic syndrome, with their associated morbidity, amongst men with locally advanced, biopsy confirmed adenocarcinoma of the prostate (PCa) that are planned to receive curative intent therapy with androgen deprivation therapy (ADT) and external beam radiotherapy (EBRT) to the prostate.

Males of any age with biopsy confirmed high tier intermediate risk PCa (Gleason score 7 and PSA 10-20) or high risk PCa (any T3; and/or Gleason Score ≥ 8.0; and/or PSA ≥ 20 ng/mL) ECOG 0 to 1, non-diabetic with no evidence of metastatic PCa will be randomized to either:

Group A: Metformin 500mg PO TID x 30-36 months total, with neoadjuvant and adjuvant ADT x18-36 months and EBRT of 46 Gy/23# to pelvic lymph nodes (optional); plus prostate boost to 78 Gy/39# or brachytherapy boost (110-115 Gy) or hypofractionated equivalent

OR

Group B: Identical placebo TID x 20-36 months total, with neoadjuvant and adjuvant ADT x18-36 months and EBRT of 46 Gy/23# to pelvic lymph nodes (optional); plus prostate boost to 78 Gy/39# or brachytherapy boost (110-115 Gy) or hypofractionated equivalent

A planned sample size of 104 patients will provide 97% power for a 2-tailed α of 0.05 to detect 4 kg difference in weight at 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Males ≥ 18 years of age
2. Pathologically confirmed, adenocarcinoma of the prostate with either high-tier intermediate or high risk prostate cancer:

   a. High-tier intermediate risk prostate cancer: i. Gleason score = 7 and PSA 10 - 20 ng/mL b. High risk prostate cancer: i. any T3; or ii. Gleason Score ≥ 8.0; or iii. PSA ≥ 20 ng/mL.
3. Normoglycemic or Impaired Fasting Glucose45 defined as:

   1. Fasting Plasma Glucose of ≤ 6.9; or
   2. HbA1c of <6.5%
4. Deemed fit to undergo curative intent external beam radiation therapy with concurrent androgen deprivation therapy by their attending radiation oncologist.
5. Accessible for follow-up clinical and laboratory assessments.

Exclusion Criteria:

1. Patients with evidence (either by imaging or pathology) of distant metastatic spread of their disease.

   a. Patients with pelvic lymph nodes (i.e. N1 disease) are NOT considered to have distant metastases and can be included in the trial, if meeting the other study criteria.
2. Patients that meet ≥1 of the Canadian Diabetes Association criteria45 for the diagnosis of diabetes:

   1. Fasting Plasma Glucose of ≥ 7.0 mmol/L; or
   2. HbA1C ≥ 6.5%; or
   3. Plasma Glucose level of ≥ 11.1 mmol/L 2 hours following a 75g oral glucose load, if known, within past 28 days; or
   4. Random Plasma Glucose level of ≥ 11.1 mmol/L, if known, within past 28 days
3. Patient who currently take metformin or those who have taken metformin within the past 12 months.
4. History of lactic acidosis or conditions that predispose to lactic acidosis including32:

   a. Impaired Renal Function (eGFR < 30); or b. Liver disease, including alcoholic liver disease, as demonstrated by any of the following parameters: i. AST >1.8 x the upper limit of normal ii. ALT > 1.8 x the upper limit of normal iii. Alkaline Phosphatase > 2x the upper limit of normal iv. Serum total bilirubin ≥ upper limit of normal c. Alcohol abuse (habitual intake of ≥3 alcoholic beverages per day) sufficient to cause hepatic toxicity d. Severe infection
5. Patients with prior bilateral orchiectomy.
6. Patients with prior prostatectomy
7. Patients who are unable to provide informed consent
8. Prior history of malignancy (with exception of adequately treated non-melanomatous skin cancer or other solid tumors treated curatively with no evidence of disease for ≥ 5 years).
9. Patients on hormonal therapy for more than 3 months prior to registration in the trial.

   -

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2014-09; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Mean body weight at 12 months of follow-up | 12 months of follow-up

SECONDARY OUTCOMES:
Prevalence and incidence of Metabolic Syndrome | At 6, 12, 24 and 36 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nawaid Usmani, MD, Principal Investigator — Cross Cancer Institute
Locations (3):
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Prairie Mountain Health - Western Manitoba Cancer Centre, Brandon, Manitoba
  - CancerCare Manitoba, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No